CLINICAL TRIAL: NCT06425484
Title: The Comparison of Effectiveness Between Epidural Combined Bilateral US TAP Block Versus Epidural Alone for Gynaecology Operation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Prof Madya, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: USM/JEPeM/kk/23010129
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Intervention Model Description: Total sample size of 46 subjects, divided into 2 groups epidural alone (Group E) and epidural with bilateral US TAP block (Group T)
Who Masked: Outcomes Assessor
Masking Description: APS team will be assessing participants pain score in the ward and documented the data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Experimental): Group epidural with bilateral US TAP block
  Interventions: Other: Bilateral US TAP block
- Group E (Active Comparator): Group epidural alone
  Interventions: Other: Bilateral US TAP block

INTERVENTIONS:
Other: Bilateral US TAP block — epidural plus bilateral US guided TAP block

SUMMARY:
The goal of this clinical trial is to compare effectiveness between epidural combined with TAP block versus epidural alone in gynaecology operation participant .The main question[s] it aims to answer are:

* what is the pain score for both groups
* what is the requirement of epidural infusion between the 2 groups Participants will be given general anesthesia for the operation with the epidural insertion prior to induction. Patient will be randomized into epidural plus TAP block or epidural alone for the study. The US TAP block will be given at the end of operation prior to extubation.

Researchers will compare pain score, epidural infusion requirment between the two groups.

DETAILED DESCRIPTION:
The research is a prospective randomized control study. It is blinded study as accessor is blinded whereby the acute pain service (APS) team will be reviewing patient postoperatively.

Study size of 46 subjects based on repeated measure ANOVA between factor , alpha value 0.05% with 80% power study, a dropout 10%. Divided into 2 groups ; Group E - epidural alone, Group T - epidural plus bilateral US TAP block.

Perioperatively, epidural catheter will be inserted then induction for general anesthesia given. Intraoperatively anesthesia maintain with inhalation agent. Prior to extubation, bilateral TAP block is provided using portable US guidance. At this location, the 3 layers of anterior abdominal wall is visualized for the truncal block. Post operatively, participant will be given epidural cocktail bupivacaine 0.1% + fentanyl 2mcg/ml infusion for next 24hrs.

The APS team will review patient post operatively in ward and all data will be recorded. Participation of patient's during study is approximately 2 days duration.

ELIGIBILITY:
Inclusion Criteria:

* Elective major laparotomy gynaecology procedure.
* Age 18 years and above
* ASA I, II, III

Exclusion Criteria:

* Prolonged INR
* Allergic to LA
* History of chronic pain
* Psychological disorder/addict to opioid or benzodiazepine
* Any contraindication for epidural or TAP block procedure
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain score between epidural plus bilateral TAP block and epidural alone | Post operatively, until day 2 post operation.
  To compare the pain score between 2 groups (epidural with bilateral TAP block) and epidural alone for gynaecology operation.

SECONDARY OUTCOMES:
To compare the epidural infusion requirement between the 2 groups ( Group T and Group E) | Post operatively, until day 2 post operation.
  To compare the postoperative epidural infusion requirement between bilateral US guided TAP block plus epidural versus epidural alone.
To evaluate time of early mobilization between 2 groups ( Group T and Group E) | Post operatively, until day 2 post operation.
  To evaluate time taken for early mobilization between group Epidural with TAP block and epidural alone after the operation .

CONTACTS AND LOCATIONS:
Overall Officials: Munirah Abdul Majid, Principal Investigator — University Sains Malaysia; W.Mohd Nazaruddin W. Hassan, Study Director — University Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganapathy S, Sondekoppam RV, Terlecki M, Brookes J, Das Adhikary S, Subramanian L. Comparison of efficacy and safety of lateral-to-medial continuous transversus abdominis plane block with thoracic epidural analgesia in patients undergoing abdominal surgery: A randomised, open-label feasibility study. Eur J Anaesthesiol. 2015 Nov;32(11):797-804. doi: 10.1097/EJA.0000000000000345. PMID 26426576
- [Background] Yoshida T, Furutani K, Watanabe Y, Ohashi N, Baba H. Analgesic efficacy of bilateral continuous transversus abdominis plane blocks using an oblique subcostal approach in patients undergoing laparotomy for gynaecological cancer: a prospective, randomized, triple-blind, placebo-controlled study. Br J Anaesth. 2016 Dec;117(6):812-820. doi: 10.1093/bja/aew339. PMID 27956680
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] Iyer SS, Bavishi H, Mohan CV, Kaur N. Comparison of Epidural Analgesia with Transversus Abdominis Plane Analgesia for Postoperative Pain Relief in Patients Undergoing Lower Abdominal Surgery: A Prospective Randomized Study. Anesth Essays Res. 2017 Jul-Sep;11(3):670-675. doi: 10.4103/0259-1162.206856. PMID 28928569
- [Result] Wu Y, Liu F, Tang H, Wang Q, Chen L, Wu H, Zhang X, Miao J, Zhu M, Hu C, Goldsworthy M, You J, Xu X. The analgesic efficacy of subcostal transversus abdominis plane block compared with thoracic epidural analgesia and intravenous opioid analgesia after radical gastrectomy. Anesth Analg. 2013 Aug;117(2):507-13. doi: 10.1213/ANE.0b013e318297fcee. Epub 2013 Jun 6. PMID 23744953
- [Result] Huepenbecker SP, Cusworth SE, Kuroki LM, Lu P, Samen CDK, Woolfolk C, Deterding R, Wan L, Helsten DL, Bottros M, Mutch DG, Powell MA, Massad LS, Thaker PH. Continuous epidural infusion in gynecologic oncology patients undergoing exploratory laparotomy: The new standard for decreased postoperative pain and opioid use. Gynecol Oncol. 2019 May;153(2):356-361. doi: 10.1016/j.ygyno.2019.02.017. Epub 2019 Feb 22. PMID 30798950